CLINICAL TRIAL: NCT07339930
Title: Phenotyping of Patients With Polycystic Ovary Syndrome (PCOS) in Alsace, France
Brief Title: Phenotyping of Patients With Polycystic Ovary Syndrome
Acronym: SOPK
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9772
Record Dates: First submitted 2026-01-05; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Polycystic Ovary Syndrome (PCOS)
Keywords: Polycystic ovary syndrome (PCOS); Polycystic Ovary; Endocrine disorder; Menstrual cycle disorders; Anti-Müllerian hormone (AMH)
MeSH Terms: conditions — Polycystic Ovary Syndrome; Endocrine System Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Polycystic ovary syndrome (PCOS) is the leading endocrine disorder of the reproductive system, affecting 10 to 13% of women of childbearing age. However, there is a significant delay in diagnosis, which may be due to considerable clinical heterogeneity and a lack of information among the general population. The diagnosis is made when two of the three Rotterdam criteria established in 2003 and revised in 2023 are met, namely: 1) menstrual cycle disorders (oligoanovulation) - 2) clinical or biological hyperandrogenism - 3) OPK morphological appearance or elevated anti-Müllerian hormone (AMH) levels, after exclusion of differential diagnoses. PCOS is a condition that carries a risk of metabolic complications and fertility problems due to dysovulation. Patients have an impaired quality of life and are at greater risk of anxiety and depression, which should be screened for systematically.

ELIGIBILITY:
Inclusion Criteria:

* Adult woman (≥18 years and <50 years)
* Subject who consulted at the Strasbourg University Hospitals for suspected PCOS or for any other endocrinological condition that led to the discovery of PCOS.

Exclusion Criteria:

* Final diagnosis excluding PCOS.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adult woman (≥18 years and <50 years) who consulted at the Strasbourg University Hospitals for suspected PCOS or for any other endocrinological condition that led to the discovery of PCOS.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09-17 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09-17 (Estimated)

PRIMARY OUTCOMES:
Prevalence of obesity | Up to 12 months
  The prevalence of obesity indicates the proportion of obese individuals in a population (a country, a region, a school, etc.) at a given time.
  It is often expressed as a percentage.
  Example:
  If, in a region of 1,000 inhabitants, 200 people are obese,
  → the prevalence of obesity is 20%.
Biological Indicators of Insulin Resistance | Up to 12 months
  Biological Indicators of Insulin Resistance:
  1. Fasting Blood Glucose (Blood Sugar) Measured after 8-12 hours of fasting. Normal: ~0.70 to 1.00 g/L (3.9-5.6 mmol/L) Abnormal: ≥1.00 g/L may suggest a disorder
  2. Fasting Insulin Indicates how much insulin the body produces at rest.
     Normal (approx.): 2 to 10 µIU/mL High: > 10-12 µIU/mL → suspected insulin resistance
  3. HOMA-IR Index (most commonly used)
  Calculated with:
  fasting blood glucose × fasting insulin ÷ 22.5 (in mmol/L)
  Common interpretation:
  < 2: normal insulin sensitivity 2-2.9: possible insulin resistance
  ≥ 3: probable insulin resistance

CONTACTS AND LOCATIONS:
Locations (1):
- ervice d'Endocrinologie, Diabétologie et Nutrition - CHU de Strasbourg - France, Strasbourg, France